CLINICAL TRIAL: NCT05460754
Title: Impact of Beef on Metabolites and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Organic Advisory and Education Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: OAEC Grant 2022
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Organic grass-fed; Conventional-fed

STUDY DESIGN:
Intervention Model Description: The design is 2 x 2 crossover design, where the healthy adults will be randomized into Organic grass-fed and conventional-fed conditions for the first round of data collection and then crossover to the other condition for the second round of data collection.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Organic grass-fed and conventional-fed steak meals were designed to be comparable in size, taste and appearance. The steaks are cut, measured in terms of size and appearance and coded prior to receipt by the research team. Randomization is for order of coded steaks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organic grass-fed beef, then conventional-fed beef (Experimental): Participants receive an organic grass-fed steak meal in the morning. After a washout period of at least 7 days, they then receive the alternative meal, conventional-fed steak meal in the morning.
  Interventions: Behavioral: Conventional-fed beef; Behavioral: Organic grass-fed beef
- Conventional-fed beef, then organic grass-fed beef (Experimental): Participants receive a conventional-fed steak meal in the morning. After a washout period of at least 7 days, they then receive the alternative meal, an organic grass-fed steak meal in the morning.
  Interventions: Behavioral: Conventional-fed beef; Behavioral: Organic grass-fed beef

INTERVENTIONS:
Behavioral: Conventional-fed beef — Participants in the conventional-fed treatment of the study will consume a conventional-fed steak meal for breakfast one morning.
Behavioral: Organic grass-fed beef — Participants in the organic grass-fed treatment of the study will consume a organic grass-fed steak meal for breakfast one morning.

SUMMARY:
Western omnivore diets tend to use beef as a good source of protein. Studies have shown cattle who are fed different diets results in varying nutritional meat profiles in terms of amino acids, types and relative amounts of fat, and other nutrients. While overlap between organic and conventionally raised beef is expected, dietary impacts on human health are potentially meaningful as small changes in diet may have large downstream effects on human metabolism. To date, no studies have been conducted in humans that evaluate the health effects of organic grass-fed beef consumption to conventionally-fed beef consumption. To fill this gap in research, the investigators propose to identify metabolic differences in response to consumption of organic grass-fed compared to conventional-fed beef on a wide array of blood borne nutrients including amino acids, lipids, bile acids, and hundreds of other metabolites. This comprehensive analysis is expected to differentiate nutritional and metabolic impacts relevant to human health and provide a foundation for future research.

The purpose of this study is to determine how a beef steak meal may affect bile acids in the gut, inflammation, and the metabolic health of healthy individuals. This research will investigate the following questions:

1. How do specific foods affect bile acids in the blood?
2. How do specific foods changes inflammation, metabolism, and other health measures? If researchers learn how food affects different health related markers in the blood and how that may influence health, then this information can be used to do more research to improve the health of people in a future study.

DETAILED DESCRIPTION:
The approach for this study is to enroll a population of healthy individuals (n=10; 5 men and 5 women) in a double-blind, two-armed (Organic Grass-fed and Conventional-fed), randomized, crossover trial in which each individual participant serves as their own control to compare postprandial serum bile acid responses between steak meals, one which is organically grass-fed (OGF) and the other conventionally-fed (CONVF). Participants will consume a 6-oz steak meal grilled to 158°F, the recommended temperature by the USDA. The randomized crossover design with half of the participants starting in the OGF arm and the other half starting in the CONVF arm will eliminate potential order effects. Block randomization with 2 blocks (total of 5 per block) will be created. Having each person serve as their own control in a crossover trial will eliminate the influence of inter-individual variation. The MSU Nutrition Research team has extensive experience with postprandial testing protocols and dietary manipulation and will utilize this experience to perform the proposed protocol with appropriate pre-test standardization, uniformity of meal preparation, precise timing of blood collection, and established procedures for processing and analyzing blood samples. Bile acids, including all primary and secondary forms, will be analyzed from samples collected before the meal and at 30-minute intervals for 4 hours after the meal. Established methods in the MSU Proteomics, Metabolomics, and Mass Spectrometry Facility will be used to compare total and individual bile acids between OGF and CONVF conditions.

Procedures:

During Visit 1, participants will undergo informed consent, be asked to complete a series of written questionnaires and anthropometric measurements. There will be a minimum 72 run-in period just prior to Visit 2, during which participants will be asked to follow certain dietary guidelines, such as no red meat. The second (Visit 2) and third (Visit 3) visits will take approximately 5 hours each and will each include a total of 9 blood draws through a sampling catheter, with each blood draw collecting about 2-3 teaspoons of blood. Blood will be drawn before a provided steak meal then every thirty minutes for 4 hours after meal consumption. There are a minimum of 72-hours between visits 1 and 2, and 7 days between visits 2 and 3. During this minimum 72- hour and 7-day period, participants will be asked to follow provided dietary and physical activity instructions. In addition, participants will be asked to complete a one month diet history questionnaire and a 24-hour dietary recall.

Dietary intervention: A meat science specialist will select and prepare the steaks which will be given to participants. Participants will be asked to consume a 6-ounce beef steak meal, cooked to 158°F that is either OGF or CONVF, but will be coded and labeled to ensure blinding.

Kinetics (measures over time) and untargeted and targeted metabolomics (an advance analytical technique to measure 1000's of molecules in a single sample) will be used as a tool to differentiate potential health impacts of the separate meal tests to investigate the influence of organic grass-fed beef versus conventionally-fed beef consumption on fasting and postprandial responses in healthy adults. The investigators expect to identify an array of metabolic differences between beef samples and will identify known impacts of those differences on health to provide a substantive comparison and provide a foundation for future research.

Metabolomic and Lipidomic analysis: When all samples have been collected, the serum samples will be thawed, and a metabolite fraction will be extracted. After extraction, the samples will be explored using mass spectrometry analysis. An initial targeted analysis will focus on bile acids, lipids, and amino acids. Targeted analytes will be quantified using standard curves and the resulting concentrations will be compared using several statistical analysis tools. Metabolite samples will be analyzed using a Waters Synapt G2Si QTOF (Waters Corporation). This instrument has ion mobility capability and can differentiate closely related compounds, such as bile acids, in complex mixtures based on their cross-sectional area and mass. The high sensitivity and variety of scan modes make the Synapt QTOF the optimal choice for untargeted analysis of complex biological samples.

Dietary analysis: This study will use the most recent version (2018) of the web-based Diet History Questionnaire (DHQ III), a food frequency questionnaire designed for adults 19 and older, developed by staff at the Risk Factor Monitoring and Methods Branch (RFMMB) of the NIH National Cancer Institute. The outputs of the DHQ III include carbohydrate constituents, carotenoids and tocopherols, dietary constituents from supplements, fats, fatty acids and cholesterol, macronutrients and energy, minerals, protein constituents, and vitamins are dietary constituents and food groups available in the DHQ III output files. In addition, acute dietary consumption will be determined using the free, web-based Automated Self-Administered 24-hour (ASA24®) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-45 years old; equal numbers male and female
* Body mass index between 18-27 kg/m^2.

Exclusion Criteria:

* Allergy to red meat
* Pregnant or Lactating
* Taking cholesterol, lipid-lowering, or anti-inflammatory medication(s)
* Antibiotic Use within the past 90 days.
* Existing gallbladder condition or gallbladder removal
* Other health concerns or conditions that may interfere with study participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Nutrition Research Laboratory, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Organic Grass-fed Beef, Then Conventional-fed Beef | Conventional-fed Beef, Then Organic Grass-fed Beef
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Organic Grass-fed Beef, Then Conventional-fed Beef | Conventional-fed Beef, Then Organic Grass-fed Beef | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (2.7) | 29 (7.31) | 26.3 (5.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Serum Lipids
Description: Concentration of postprandial serum triglycerides, high-density lipoproteins, cholesterol (mM)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Organic Grass-fed Beef: Participants receive an organic grass-fed steak meal in the morning. After a washout period of at least 7 days, they then receive the alternative meal, conventional-fed steak meal in the morning.
  Organic grass-fed beef: Participants in the organic grass-fed treatment of the study will consume a organic grass-fed steak meal for breakfast one morning.
- Conventional-fed Beef: Participants receive a conventional-fed steak meal in the morning. After a washout period of at least 7 days, they then receive the alternative meal, an organic grass-fed steak meal in the morning.
  Conventional-fed beef: Participants in the conventional-fed treatment of the study will consume a conventional-fed steak meal for breakfast one morning.
Arm/Group | Organic Grass-fed Beef | Conventional-fed Beef
Number analyzed (Participants) | 10 | 10
mmol/L
  Triglycerides Hour 0 | 1.01 (0.48) | 0.94 (0.43)
  Triglycerides Hour 1 | 0.99 (0.52) | 0.97 (0.43)
  Triglycerides Hour 2 | 1.009 (0.53) | 1.09 (0.48)
  Triglycerides Hour 3 | 1.14 (0.61) | 1.27 (0.71)
  Triglycerides Hour 4 | 1.16 (0.62) | 1.26 (0.69)
  HDL Hour 0 | 1.46 (0.21) | 1.38 (0.16)
  HDL Hour 1 | 1.45 (0.16) | 1.41 (0.17)
  HDL Hour 2 | 1.46 (0.23) | 1.38 (0.13)
  HDL Hour 3 | 1.46 (0.19) | 1.39 (0.17)
  HDL Hour 4 | 1.45 (0.21) | 1.37 (0.16)
  Cholesterol Hour 0 | 3.92 (1.04) | 3.74 (0.76)
  Cholesterol Hour 1 | 3.97 (1.023) | 3.84 (0.80)
  Cholesterol Hour 2 | 3.97 (1.08) | 3.81 (0.85)
  Cholesterol Hour 3 | 3.97 (1.06) | 3.84 (0.79)
  Cholesterol Hour 4 | 3.85 (1.06) | 3.84 (0.78)

2. Secondary Outcome: Postprandial Serum Inflammatory Cytokines
Description: Concentration of postprandial serum inflammatory cytokine responses (tumor necrosis factor-alpha, interleukin-(IL)1beta, IL-6, IL-10, IL-17, IL-23, interferon-gamma, and granulocyte macrophage-colony stimulating factor; all in pg/ml)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Organic Grass-fed Beef | Conventional-fed Beef
Number analyzed (Participants) | 10 | 10
pg/ml
  TNFa Hour 0 | 17.84 (5.57) | 17.65 (5.92)
  TNFa Hour 1 | 17.62 (5.37) | 17.69 (6.12)
  TNFa Hour 2 | 18.35 (6.38) | 17.27 (5.29)
  TNFa Hour 3 | 17.14 (5.57) | 17.87 (5.90)
  TNFa Hour 4 | 17.08 (7.21) | 17.59 (7.82)
  IL-1b Hour 0 | 6.64 (2.07) | 6.89 (2.08)
  IL-1b Hour 1 | 6.76 (1.80) | 6.69 (2.31)
  IL-1b Hour 2 | 6.8 (1.93) | 6.70 (2.40)
  IL-1b Hour 3 | 6.7 (2.35) | 6.64 (2.25)
  IL-1b Hour 4 | 6.84 (3.21) | 6.93 (2.74)
  IL-6 Hour 0 | 7.55 (9.24) | 7.69 (11.00)
  IL-6 Hour 1 | 8.44 (9.98) | 7.47 (10.18)
  IL-6 Hour 2 | 8.73 (11.46) | 6.90 (7.41)
  IL-6 Hour 3 | 8.38 (11.76) | 8.44 (11.47)
  IL-6 Hour 4 | 6.87 (7.91) | 8.07 (11.10)
  IL-10 Hour 0 | 71.55 (45.54) | 72.67 (54.50)
  IL-10 Hour 1 | 76.79 (52.01) | 73.28 (52.87)
  IL-10 Hour 2 | 79.11 (58.30) | 72.56 (51.45)
  IL-10 Hour 3 | 73.83 (57.94) | 76.40 (60.46)
  IL-10 Hour 4 | 67.50 (58.54) | 74.45 (59.98)
  IL-17 Hour 0 | 76.02 (31.58) | 77.59 (36.29)
  IL-17 Hour 1 | 80.16 (33.65) | 81.01 (44.62)
  IL-17 Hour 2 | 82.41 (40.20) | 78.43 (31.96)
  IL-17 Hour 3 | 74.20 (34.27) | 86.14 (39.63)
  IL-17 Hour 4 | 73.59 (40.40) | 85.76 (44.09)
  IL-23 Hour 0 | 957.70 (402.55) | 1020.18 (571.19)
  IL-23 Hour 1 | 989.14 (434.31) | 1051.23 (614.26)
  IL-23 Hour 2 | 1042.90 (549.85) | 1039.69 (473.53)
  IL-23 Hour 3 | 949.10 (517.76) | 1045.52 (547.79)
  IL-23 Hour 4 | 917.97 (646.34) | 1037.87 (658.14)
  INF Hour 0 | 343.49 (232.40) | 363.51 (258.16)
  INF Hour 1 | 376.34 (264.81) | 402.29 (318.26)
  INF Hour 2 | 391.97 (298.69) | 357.08 (214.32)
  INF Hour 3 | 354.88 (249.63) | 399.32 (287.39)
  INF Hour 4 | 375.96 (282.53) | 405.13 (316.27)
  GMCSF Hour 0 | 67.14 (38.25) | 64.29 (37.73)
  GMCSF Hour 1 | 61.46 (34.62) | 59.62 (33.01)
  GMCSF Hour 2 | 58.72 (30.09) | 59.76 (35.88)
  GMCSF Hour 3 | 57.47 (32.08) | 60.98 (32.21)
  GMCSF Hour 4 | 58.86 (38.67) | 61.99 (34.27)

3. Secondary Outcome: Postprandial Serum Glucose
Description: Serum glucose concentration (mM)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Organic Grass-fed Beef | Conventional-fed Beef
Number analyzed (Participants) | 10 | 10
mmol/L
  Hour 0 | 5.52 (0.86) | 5.41 (0.81)
  Hour 1 | 5.19 (0.69) | 5.06 (0.76)
  Hour 2 | 5.21 (0.63) | 5.17 (0.72)
  Hour 3 | 5.38 (0.82) | 5.34 (0.86)
  Hour 4 | 5.44 (0.74) | 5.37 (0.72)

4. Secondary Outcome: Postprandial Serum Insulin
Description: Serum insulin concentration (microIU/mL)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: microIU/mL
Arm/Group | Organic Grass-fed Beef | Conventional-fed Beef
Number analyzed (Participants) | 10 | 10
microIU/mL
  Hour 0 | 8.99 (7.48) | 6.28 (3.92)
  Hour 1 | 13.95 (9.20) | 15.08 (8.29)
  Hour 2 | 12.60 (7.68) | 12.307 (8.65)
  Hour 3 | 16.28 (29.04) | 8.95 (5.94)
  Hour 4 | 9.97 (18.19) | 9.58 (10.10)

ADVERSE EVENTS:
Time Frame: 0 months
Description: We did not collect adverse events data after the participant complete the study
Arm/Group | Organic Grass-fed Beef | Conventional-fed Beef
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT05460754/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT05460754/SAP_001.pdf
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT05460754/ICF_002.pdf